CLINICAL TRIAL: NCT04246775
Title: Low Anterior Resection Syndrome and Rectal Irrigation Study
Acronym: LARRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: South East Wales Trials Unit (SEWTU) (Unknown); Tenovus (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIHR/UKCRN Portfolio ID: 18113
Record Dates: First submitted 2015-02-10; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2015-02

CONDITIONS: Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Peristeen given
  Interventions: Device: Peristeen

INTERVENTIONS:
Device: Peristeen — rectal irrigation

SUMMARY:
Prospective study assessing treatment acceptability and the impact of rectal irrigation on patients with low anterior resection syndrome (LARS) in terms of quality of life and bowel function.

DETAILED DESCRIPTION:
Aims: To assess if rectal irrigation improves patient symptoms and quality of life in patients with LARS and to see if the treatment is acceptable to patients.

Methods: This is a mixed methods evaluation study on functional outcomes in patients who have undergone anterior resection for rectal neoplasia and who have had bowel continuity restored between Jan 2009 and Jan 2014. Those patients deemed to have LARS who consent to participation in the study will be offered rectal irrigation.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone anterior resection for rectal neoplasia, patients who have had restored bowel continuity
* LARS score of >20 (defined LARS syndrome)
* patients > 18 years of age.

Exclusion Criteria:

* previous use of rectal irrigation
* patients who are unable to give informed consent
* patients who are not physically capable of performing the treatment in their home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
SF12 | pre intervention and 6 months post
  quality of life

SECONDARY OUTCOMES:
EORTC | pre intervention and 6 months post
  quality of life
Low anterior resection score | pre intervention and 6 months post
  bowel function
St Marks Faecal incontinence score | pre intervention and 6 months post
  bowel function
treatment acceptability questionnaire | post training for treatment and 6 months post treatment

OTHER OUTCOMES:
qualitative interviews | after 6 months treatment or drop out from treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom